CLINICAL TRIAL: NCT01081158
Title: Assessment of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SCH 900518 in Naive or Treatment-Experienced Subjects Infected With Hepatitis C Virus Genotype 1 (Protocol No. P04695)
Brief Title: Safety, Tolerability, PK and PD of SCH 900518 in Naive or Treatment-Experienced Subjects Infected With HCV Genotype 1 (Protocol No. P04695)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04695
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — narlaprevir; peginterferon alfa-2b; Ritonavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment-naïve 800 mg TID (Experimental): Period 1: SCH 900518 (800 mg TID) or placebo for 7 days
  Period 2: SCH 900518 (800 mg TID) + PegIntron (1.5 µg/kg QW) or placebo + PegIntron for 14 days.
  Interventions: Drug: Drug: SCH 900518 Biologic: Peginterferon alfa-2b(PegIntron)
- Treatment-experienced: 800 mg TID (Experimental): Period 1: SCH 900518 (800 mg TID) or placebo for 7 days
  Period 2: SCH 900518 (800 mg TID) + PegIntron (1.5 ug/kg QW) or placebo + PegIntron for 14 days
  Interventions: Drug: Drug: SCH 900518 Biologic: Peginterferon alfa-2b
- Treatment-naïve: 400 mg + RTV BID (Experimental): Period 1: SCH 900518 (400 mg BID) or placebo + RTV (200 mg BID) for 7 days.
  Period 2: SCH 900518 (400 mg BID) or placebo + RTV (200 mg BID) +PegIntron (1.5 µg/kg QW) for 14 days.
  Interventions: Drug: Drug: SCH 900518 Drug: Ritonavir (RTV) Biologic: Peginterferon alfa-2b (PegIntron)
- Treatment-experienced: 400 mg + RTV BID (Experimental): Period 1: SCH 900518 (400 mg BID) or placebo + RTV (200 mg BID) for 7 days.
  Period 2: SCH 900518 (400 mg BID) or placebo + RTV (200 mg BID) +PegIntron (1.5 µg/kg QW) for 14 days.
  Interventions: Drug: Drug: SCH 900518 Drug: Ritonavir (RTV) Drug: Ritonavir (RTV) Biologic: Peginterferon alfa-2b (PegIntron)

INTERVENTIONS:
Drug: Drug: SCH 900518 Biologic: Peginterferon alfa-2b(PegIntron) — Drug: SCH 900518
  Biologic: Peginterferon alfa-2b(PegIntron)
  Period 1: Amorphous SCH 900518 800 mg or placebo TID administered as an oral suspension for 7 days .
  Period 2: Amorphous SCH 900518 800 mg or placebo TID administered as an oral suspension for 14 days in combination with 1.5 µg/kg PegIntron administered subcutaneously weekly.
  Other Names: narlaprevir, PegIntron
  Arms: Treatment-naïve 800 mg TID
Drug: Drug: SCH 900518 Biologic: Peginterferon alfa-2b — Drug: SCH 900518
  Biologic: Peginterferon alfa-2b
  Period 1: Amorphous SCH 900518 800 mg or placebo TID administered as an oral suspension for 7 days
  Period 2: Amorphous SCH 900518 800 mg or placebo TID administered as an oral suspension for 14 days in combination with 1.5 µg/kg PegIntron administered subcutaneously weekly.
  Other Names: narlaprevir, PegIntron
  Arms: Treatment-experienced: 800 mg TID
Drug: Drug: SCH 900518 Drug: Ritonavir (RTV) Biologic: Peginterferon alfa-2b (PegIntron) — Drug: SCH 900518
  Drug: Ritonavir (RTV)
  Biologic: Peginterferon alfa-2b (PegIntron)
  Period 1: Amorphous SCH 900518 (400 mg) or placebo BID administered as oral suspension + ritonavir (200 mg BID) (2-100 mg oral capsules) for 7 days.
  Period 2: Amorphous SCH 900518 (400 mg) or placebo BID administered as oral suspension+ ritonavir (200 mg BID) (2-100 mg oral capsules) + PegIntron (1.5 µg/kg QW) for 14 days.
  Other Names: narlaprevir, norvir, PegIntron
  Arms: Treatment-naïve: 400 mg + RTV BID
Drug: Drug: SCH 900518 Drug: Ritonavir (RTV) Drug: Ritonavir (RTV) Biologic: Peginterferon alfa-2b (PegIntron) — Drug: SCH 900518
  Drug: Ritonavir (RTV)
  Biologic: Peginterferon alfa-2b (PegIntron)
  Period 1, Amorphous SCH 900518 (400 mg) or placebo BID administered as an oral suspension + RTV (200 mg BID) oral capsules (2-100 mg capsules) for 7 days.
  Period 2, SCH 900518 (400 mg) or placebo BID as an oral suspension + RTV (200 mg BID) oral capsules (2-100 mg capsules) +PegIntron (1.5 µg/kg SC QW) for 14 days.
  Other Names: narlaprevir, norvir, PegIntron
  Arms: Treatment-experienced: 400 mg + RTV BID

SUMMARY:
Assessment of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SCH 900518 in Naive or Treatment-Experienced Subjects Infected With Hepatitis C Virus Genotype 1 (Protocol No. P04695)

ELIGIBILITY:
Inclusion Criteria:

* Subject infected with HCV genotype 1 (any sub-type) virus who is:

  * treatment naïve (eg. to interferon and ribavirin); or
  * treatment experienced (non-responder and relapser): subject who received interferon based therapy and continued to have detectable HCV RNA levels at the end of follow-up, a subject who did not attain a 2 log decline in HCV RNA levels at ~12 weeks and discontinued treatment, or subject who had no detectable viral load while on treatment but had a detectable viral load post treatment.
* Subject with acceptable medical history, physical examination, and clinical laboratory evaluations consistent with CHC, compensated liver disease, and any associated diseases (diabetes, hypertension, etc).
* Subjects with an HCV RNA viral load of >10^5 copies/mL or equivalent international units

BMI of 18 to 40 kg/m^2, men and women, ages 18-65 years inclusive

* Female must be non-lactating and have a negative pregnancy test at Screening and Day -1 and either be of nonchildbearing potential or if of childbearing potential, must be practicing effective double-barrier contraceptive methods from at least 2 weeks prior to Day -1 until 30 days after study completion.
* Male must be willing to practice barrier contraception from Day 1 through 3 months following treatment with SCH 900518.
* Subject must have an ECG recording showing no clinically significant findings at Screening.
* Subject with chronic stable hemophilia may enroll
* Subject on stable methadone treatment may enroll in this study (evaluation by investigator includes history of stable clinical management for >3 months).

Exclusion Criteria:

* Subject has a significant acute or chronic medical illness which is not stable or is not controlled with medication (excluding prohibited medications).
* Subject has received an organ transplant.
* Subject has evidence of decompensated liver disease by physical exam (encephalopathy, ascites, caput medusae, etc).
* Subject has at anytime received an HCV NS3-specific protease inhibitor.
* Subject has a platelet count <80,000/mm^3 (confirmed by repeat analysis) at Screening.
* Subject has a serum hemoglobin of <10.0 g/dL (confirmed by repeat analysis) at Screening.
* Subject has a serum AST /ALT value >5 x ULN (confirmed by repeat analysis) at Screening.
* Subject has a serum alkaline phosphatase value >2 x ULN (confirmed by repeat analysis) at Screening.
* Two or more of the following criteria (confirmed by repeat analysis) at Screening:

  * Total serum bilirubin >2.0 mg/dL.
  * Serum albumin <3.5 g/dL.
  * INR >1.7 (with the exception of hemophiliacs).
* Subject has a neutrophil count <1,000/mm^3 (confirmed by repeat analysis) at Screening.
* Creatinine clearance (as estimated by method of Cockcroft and Gault) less than 50 mL/min at Screening.
* Subject who has a history of any clinically significant local or systemic infectious disease within 1 week prior to screening (other than HCV-infection).
* Male subject whose female partner intends on becoming pregnant within 3 months of the study.
* Subject is positive for HIV antibodies or hepatitis B surface antigen.
* Subject has a clinically significant allergy or intolerance to foods or drugs, or is known or suspected to have hypersensitivity to any ingredient in the investigational product.
* Subject has a clinically significant history of auto-immune hepatitis.
* Subject has used any investigational drugs or donated blood within 30 days prior to study drug administration.
* Subject who received any of the following treatments: known inhibitor of CYP3A4 metabolism (2 weeks of prior to randomization), known inducer of CYP3A4 metabolism (2 weeks prior to randomization) and treatment for HCV infection (1 month prior to randomization)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability were to be assessed by collecting adverse events (AEs), vital signs, electrocardiograms (ECGs), physical examinations, urinalysis, and safety laboratory tests. | Screening Period: 90 days, Period 1: 7 days, Washout: 4 weeks, Period 2: 14 days, Standard of Care with PegIntron and ribavirin: 84 days

SECONDARY OUTCOMES:
Log change in HCV-RNA from baseline. Ctrough of SCH 900518 resulting in mean HCV RNA decrease > 2 log10 IU/mL. Ctrough of SCH 900518+PEG resulting in HCV-RNA < LOQ. SCH 900518 PK: Cmax, Tmax, AUC, Ctrough, t½, R, CL/F, Vd/F. PEG and RTV: Ctrough | Period 1: 7 days, Washout: 4 weeks, Period 2: 14 Days

REFERENCES:
- [Result] de Bruijne J, Bergmann JF, Reesink HW, Weegink CJ, Molenkamp R, Schinkel J, Tong X, Li J, Treitel MA, Hughes EA, van Lier JJ, van Vliet AA, Janssen HL, de Knegt RJ. Antiviral activity of narlaprevir combined with ritonavir and pegylated interferon in chronic hepatitis C patients. Hepatology. 2010 Nov;52(5):1590-9. doi: 10.1002/hep.23899. PMID 20938912
- [Result] Hotho DM, de Bruijne J, Spaan M, Treitel MA, Boonstra A, de Knegt RJ, Janssen HL, Reesink HW. Sustained virologic response after therapy with the HCV protease inhibitor narlaprevir in combination with peginterferon and ribavirin is durable through long-term follow-up. J Viral Hepat. 2013 Apr;20(4):e78-81. doi: 10.1111/jvh.12012. Epub 2013 Jan 7. PMID 23490393